CLINICAL TRIAL: NCT02298426
Title: Body Constitution Classification Based Comprehensive Health Management Intervention on Obese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hai-Jun Wang (Other)
Responsible Party: Sponsor-Investigator, Hai-Jun Wang, professor, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00001052-13086
Record Dates: First submitted 2014-11-09; First posted 2014-11-24 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Overweight; Obesity
Keywords: Body Constitution Classification; Health Management; Obese Population
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- health management and product (Experimental): We provide large scales of weight management information included recipes according to people's constitution. Information is provide through both face to face meeting and telephones. Materials are also given to participants.
  Meanwhile, we use dietary supplement products of "SCHSANDRA PLUS", "YI RUI CAPSULE", "Gest Aid Plus": "INFINITUS®" to help balance the constitution of participants.
  Interventions: Behavioral: Health Management; Dietary Supplement: SCHSANDRA PLUS, YI RUI CAPSULE, Gest Aid Plus: INFINITUS®
- general management and product (Experimental): We provide general information about health. Information is provided through telephones and materials.
  Meanwhile, we use dietary supplement products of "SCHSANDRA PLUS", "YI RUI CAPSULE", "Gest Aid Plus": "INFINITUS®" to help balance the constitution of participants.
  Interventions: Behavioral: General Management; Dietary Supplement: SCHSANDRA PLUS, YI RUI CAPSULE, Gest Aid Plus: INFINITUS®
- health management and placebo (Experimental): We provide large scales of weight management information included recipes according to people's constitution. Information is provide through both face to face meeting and telephones. Materials are also given to participants.
  Meanwhile, we use placebo to replace the dietary supplement products.
  Interventions: Behavioral: Health Management; Other: Placebo
- general management and placebo (Placebo Comparator): We provide general information about health. Information is provided through telephones and materials.
  Meanwhile, we use placebo to replace the dietary supplement products.
  Interventions: Behavioral: General Management; Other: Placebo

INTERVENTIONS:
Behavioral: Health Management — We provide large scales of weight management information included recipes according to people's constitution. Information is provide through both face to face meeting and telephones. Materials are also given to participants.
  Arms: health management and placebo; health management and product
Behavioral: General Management — We provide general information about health. Information is provided through telephones and materials.
  Arms: general management and placebo; general management and product
Other: Placebo — We use placebo to replace the health product.
  Arms: general management and placebo; health management and placebo
Dietary Supplement: SCHSANDRA PLUS, YI RUI CAPSULE, Gest Aid Plus: INFINITUS® — We use dietary supplement products to help balance the constitution of participants. Each participant got one of the three dietary supplement products. SCHSANDRA PLUS, INFINITUS® is a health product made of Schisandra, ginseng, Ginseng, Radix and other plant materials which can help enhance the body's antioxidant capacity. YI RUI CAPSULE , INFINITUS® is a health product made of salvia, hawthorn, alisma, perilla oil microcapsules, panax powder, ginkgo biloba and other plant materials which can assist lower the blood lipid level. Gest Aid Plus, INFINITUS® is a health product made of yam, codonopsis, poria, white beans, dried tangerine peel and other plant materials which can help regulate intestinal flora.
  Arms: general management and product; health management and product

SUMMARY:
This study aims to explore the effectiveness of body constitution classification based comprehensive health management intervention on obese population.

DETAILED DESCRIPTION:
This study aims to explore the effectiveness of body constitution classification based comprehensive health management intervention on obese population, compare the differences in effectiveness between body constitution classification based management vs usual health management, and explore the influence of different food composition on the effectiveness of body constitution classification based comprehensive health management intervention on obese population.

ELIGIBILITY:
Inclusion Criteria:

* Social characteristics:

  * 20-55 year old,
  * had lived in a city for more than one year,
  * kept a watchful eye on losing weight or bodybuilding,
  * practitioner engaged in non- sensitive sectors.
* Physiological characteristics:

  * met the obesity diagnostic criteria suggested by "Prevention and control Guidelines for overweight and obesity of Chinese adults in 2006". Subjects with a BMI between 24 to 28 kg/m2 were defined as overweight, while those with a BMI greater than 28kg/m2 were obese.
  * met the constitution classification standards of Traditional Chinese Medicine. According to the constitution questionnaire formulated on the base of the Chinese Medical Association standard "Chinese constitution classification and determination" (ZYYXH/T157-2009), the subjects were divided into phlegm-damp type, qi deficiency type and phlegm stasis block type.

Exclusion Criteria:

* with the following major organic disease,
* secondary obesity caused by diseases,
* none of phlegm-damp type, qi deficiency type or phlegm stasis block type,
* women who were planning to become pregnant, pregnant or lactating.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1452 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
BMI | Baseline,1year
  We measure the body mass index to examine the effect of weight loss Content 10% effective loss of weight Less than 15% safe loss of weight Ensure 5% loss of weight,Content 10% effective loss of weight,Less than 15% safe loss of weight

SECONDARY OUTCOMES:
Body fat percentage | Baseline,1year
  We measure the body fat percentage to examine the effect of weight loss on body composition.
Fatty liver | Baseline,1year
  We examine if the participants suffer fatty liver using the method of ultrasonic.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, Principal Investigator — Peking University
Locations (1):
- Peking University Health Science Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No